CLINICAL TRIAL: NCT01248221
Title: [13C]-Spirulina Platensis GEBT - Dual-Label Validation Study
Brief Title: Carbon-13 (13C)-Spirulina Platensis Gastric Emptying Breath Test (GEBT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH); Advanced Breath Diagnostics, LLC (Unknown)
Responsible Party: Adil E. Bharucha, M.B.B.S, M.D., Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-006643; P01DK068055 (NIH); UL1RR024150 (NIH)
Record Dates: First submitted 2010-11-23; First posted 2010-11-25 (Estimated); Results first posted 2013-03-18 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-02

CONDITIONS: Dyspepsia
Keywords: Breath test; Dyspepsia; Gastric Emptying; Gastroparesis
MeSH Terms: conditions — Dyspepsia; Gastroparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy subjects (Experimental): The subject will consume the test meal containing [13C]-Spirulina platensis and 99mTc sulfur colloid, after which gastric emptying will be assessed simultaneously by scintigraphy and breath tests. Scintigraphic image acquisition will be obtained upon completion of the meal and at 15, 30, 45, 60, 90, 120, 150, 180, and 240 minute time points. Breath samples will be collected at baseline before the test meal is started and thereafter on the same time schedule as the scintigraphic procedure.
  Interventions: Drug: [13C]-Spirulina platensis and 99mTc sulfur colloid
- Dyspeptic subjects (Experimental): The subject will consume the test meal containing [13C]-Spirulina platensis and 99mTc sulfur colloid, after which gastric emptying will be assessed simultaneously by scintigraphy and breath tests. Scintigraphic image acquisition will be obtained upon completion of the meal and at 15, 30, 45, 60, 90, 120, 150, 180, and 240 minute time points. Breath samples will be collected at baseline before the test meal is started and thereafter on the same time schedule as the scintigraphic procedure.
  Interventions: Drug: [13C]-Spirulina platensis and 99mTc sulfur colloid

INTERVENTIONS:
Drug: [13C]-Spirulina platensis and 99mTc sulfur colloid — The subject will consume the test meal containing 13C-Spirulina and 99mTc sulfur colloid in no more than 10 minutes. Scintigraphic image acquisition will be obtained upon completion of the meal and at 15, 30, 45, 60, 90, 120, 150, 180, and 240 minute time points. Breath samples will be collected at baseline before the test meal is started and thereafter on the same time schedule as the scintigraphic procedure.

SUMMARY:
The purpose of this study is to compare stomach emptying using 13C-Spirulina platensis breath test and scintigraphy in healthy subjects and subjects with dyspepsia.

Subjects will eat a standard meal of 2 scrambled eggs, a slice of wheat toast and 8 ounces of skim milk. The eggs will be double labeled with Technetium-99m (99mTc) sulfur colloid and 13C-Spirulina platensis.

Scintigraphy is a diagnostic technique in which a two-dimensional picture of internal body tissue is produced through the detection of radiation emitted by a radioactive substance administered into the body. The location of a standard meal in the digestive system will be measured by images of the 99mTc sulfur colloid taken at periodic intervals before and after the standard meal. The 99mTc Sulfur Colloid is approved by the FDA for use in medical diagnostic procedures.

Spirulina platensis is blue - green algae, which is very similar to the naturally occurring spirulina sold in health food stores as a dietary supplement. The spirulina platensis has been labeled with the 13C stable isotope. 13C stable isotope labeling is inherently safe as 1.1% of all carbon in our bodies and in the food we eat is 13C. The presence of the 13C will be measured by breath samples at periodic intervals before and after a standard meal. The FDA considers 13C-Spirulina platensis to be investigational for the purposes of this study.

DETAILED DESCRIPTION:
The objective of this study is to compare gastric emptying assessed by the modified 13C spirulina breath test and scintigraphy in 30 subjects, i.e., 15 healthy subjects and 15 with dyspepsia. Gastric emptying will be simultaneously assessed by both methods using a dual-labeled meal. It is anticipated that the gastric emptying half-time (t½) values based on the 13C breath excretion values will compare with the gold standard, scintigraphy, in which the "true" t½ values are obtained. The aims of this study are to estimate factors necessary for converting exhaled 13C concentrations to gastric emptying half-time, as measured by scintigraphy, in healthy subjects and patients with dyspepsia.

For each potential participant, a screening visit will be conducted within 4 weeks prior to the study visit. During the screening visit, informed consent will be obtained, and a physical exam will be conducted by a trained investigator. Participants will then be free to leave the test site. A urine pregnancy test for women of child-bearing potential will be completed within 48 hours prior to exposure to radiation. After an overnight (minimum 8 hour) fast, the participants will return to the study center, at which time the dual-label Gastric Emptying Test will be administered. A baseline breath sample will be collected in duplicate by having the subject blow through a straw into a collection tube. The test meal will be prepared by personnel at the test site after the subject arrives. Step-by-step test meal preparation instructions are provided with the GEBT kit. The patient will consume the test meal containing [13C]-Spirulina and 99mTc sulfur colloid in no more than 10 minutes. Scintigraphic image acquisition will be obtained upon completion of the meal and at 15, 30, 45, 60, 90, 120, 150, 180, and 240 minute time points. Breath samples will be collected at baseline before the test meal is started and thereafter on the same time schedule as the scintigraphic procedure.

As the cooked egg is triturated by the stomach, it passes through the pylorus into the intestine where the [13C]-Spirulina platensis is digested, absorbed, and metabolized giving rise to labeled carbon dioxide expired in the breath. Breath samples, collected before and after the test meal, are shipped overnight to Advanced Breath Diagnostics for analysis by Gas Isotope Ratio Mass Spectroscopy. By measuring the change in excretion over time, the rate of gastric emptying can be determined.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant, non-breastfeeding female volunteers
* 18-70 years of age
* Able to provide written informed consent before participating in the study
* Able to communicate adequately with the Investigator and to comply with the requirements of for the entire study, i.e., able to eat test meal and provide breath samples.

Additional inclusion criteria for dyspepsia patients:

* One or more of eight postprandial dyspeptic symptoms i.e., fullness, bloating, epigastric discomfort, early satiety, nausea, vomiting, belching, pain for a minimum of 3 months, OR
* Patients fulfilling the ROME-III criteria for functional dyspepsia,
* AND no symptom improvement under a standard dose proton-pump inhibitor (PPI) treatment,
* AND an upper gastrointestinal endoscopy negative for significant pathology that would explain symptoms done within the last 5 years prior to the study.

Exclusion Criteria:

* Severe nausea or vomiting precluding study assessments
* Use of medications that alter GI motility e.g., narcotics or medications with significant anticholinergic effects within two days of the study
* History of malabsorption due to mucosal disease, pancreatic disease, liver dysfunction, or other causes
* Abdominal surgery other than appendectomy, cholecystectomy, tubal ligation or hysterectomy
* Clinical evidence of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological, psychiatric, or other disease that may interfere with the objectives of the study
* Patients who are allergic to eggs, wheat, or milk, or unwilling to consume these products
* Patients who have taken any investigational medications within the past 30 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adil E Bharucha, MBBS, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from public advertisement and the motility clinic at the Mayo Clinic in Rochester, Minnesota.
Period: Overall Study
Arm/Group | Healthy Subjects | Dyspeptic Subjects
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dyspeptic Subjects | Healthy Subjects | Total
Number analyzed (Participants) | 15 | 15 | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 41.08 (14.90) | 42.01 (14.46) | 41.54 (14.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.75 (8.0) | 27.21 (6.0) | 26.98 (6.95)

OUTCOME MEASURES:

1. Primary Outcome: Gastric Emptying Half Time Measured by Scintigraphy
Description: Gastric emptying half time is the time for half of the ingested solids to leave the stomach. This value was measured by standard 99m Tc scintigraphy.
Time Frame: 4 hours after ingestion of standard meal
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Healthy Subjects; Dyspeptic Subjects: The subject will consume the test meal containing [13C]-Spirulina platensis and Technetium-99m (99mTc) sulfur colloid, after which gastric emptying will be assessed simultaneously by scintigraphy and breath tests. Scintigraphic image acquisition will be obtained upon completion of the meal and at 15, 30, 45, 60, 90, 120, 150, 180, and 240 minute time points. Breath samples will be collected at baseline before the test meal is started and thereafter on the same time schedule as the scintigraphic procedure.
Arm/Group | Healthy Subjects | Dyspeptic Subjects
Number analyzed (Participants) | 15 | 15
minutes | 65.9 (14.7) | 82.2 (34.6)

2. Primary Outcome: Gastric Emptying Half Time Measured by 13C Spirulina Gastric Emptying Breath Test (GEBT)
Description: Gastric emptying half time is the time for half of the ingested solids to leave the stomach. This value was measured by the 13C spirulina GEBT.
Time Frame: 4 hours after ingestion of standard meal
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Healthy Subjects | Dyspeptic Subjects
Number analyzed (Participants) | 15 | 15
minutes | 67.3 (14.0) | 82.5 (33.2)

3. Secondary Outcome: Gastric Emptying at 60, 120, and 240 Minutes Measured by Scintigraphy
Description: The scintigraphic gastric emptying (GE) metric is the proportion of tracer emptied from the stomach at time, t.
Time Frame: 60, 120, and 240 minutes after ingestion of standard meal
Measure: Mean (Standard Deviation); unit: proportion of tracer
Arm/Group | Healthy Subjects | Dyspeptic Subjects
Number analyzed (Participants) | 15 | 15
proportion of tracer
  GE 60 minutes | 0.467 (0.096) | 0.318 (0.137)
  GE 120 minutes | 0.784 (0.100) | 0.545 (0.164)
  GE 240 minutes | 0.978 (0.083) | 0.844 (0.167)

4. Secondary Outcome: Gastric Emptying at 60, 120, and 240 Minutes Measured by 13C Spirulina Gastric Emptying Breath Test (GEBT)
Description: A multiple linear regression model approach was used to estimate gastric emptying based on the breath test samples at each time point. Gastric emptying (GE) metric is the proportion of tracer emptied from the stomach at time, t.
Time Frame: 60, 120, and 240 minutes after ingestion of standard meal
Measure: Mean (Standard Deviation); unit: proportion of tracer
Arm/Group | Healthy Subjects | Dyspeptic Subjects
Number analyzed (Participants) | 15 | 15
proportion of tracer
  GE 60 minutes | 0.459 (0.103) | 0.324 (0.131)
  GE 120 minutes | 0.775 (0.111) | 0.556 (0.158)
  GE 240 minutes | 0.958 (0.047) | 0.847 (0.142)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the time the subjects were on the study, approximately one month.
Arm/Group | Healthy Subjects | Dyspeptic Subjects
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No